CLINICAL TRIAL: NCT07018102
Title: Nurse-Led Bedside Trunk Control Care Program for Patients With Stroke
Brief Title: Nurse-Led Bedside Trunk Control Care Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Hsiang Chu Pai, professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CS1-23077
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: trunk impairment; diaphragmatic breathing; quality of life; respiration function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trunk Control Care Program (Experimental): A step-wise nurse-led bedside trunk control care module intervention
  Interventions: Other: Trunk Control Care Program
- standard care (No Intervention): The control group received routine care including health education on turning over, positioning, and wheelchair use.

INTERVENTIONS:
Other: Trunk Control Care Program — 1. The intervention group underwent a 4-week bedside trunk control care module intervention based on routine care in a rehabilitation ward.
  2. trunk control care module: combine the care strategies of "arm training, butterfly technique, shoulder control, diaphragmatic breathing" and "body awareness", practice twice a day, each time for 20-30 minutes, and can be adjusted according to the patient's condition.
  Arms: Trunk Control Care Program

SUMMARY:
This study aimed to apply care for stroke survivors by establishing trustable professional activities competency indicators and a trunk control care module for rehabilitation ward nurses during our second year.

DETAILED DESCRIPTION:
Thus, the purposes of this study were: (1) to evaluate the effect of a stepwise nurse-led bedside trunk control care module intervention on improving trunk control, respiratory function, and quality of life in patients with stroke and (2) to modify and confirm the milestones and trustable professional activities of competence in trunk impairment care for patients with stroke to provide evidence-based nursing education and cultivate new nurses' competence in trunk injury care in the future.

ELIGIBILITY:
Inclusion Criteria:

* (a) Patients hospitalized for stroke in rehabilitation or neurology wards, currently in stable condition; (b) Trunk Impairment Scale score below 21; (c) aged 20 or above; (d) patients willing to participate.

Exclusion Criteria:

* Patients with Trunk Impairment Scale score above 21, as this indicates that they can perform daily activities independently

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Trunk function | Questionnaire were filled out three times, before the program intervention and at the two and fourth weeks following the intervention.
  Trunk Impairment Scale is used to assess patients' trunk function.

SECONDARY OUTCOMES:
Postural control | Questionnaire were filled out three times, before the program intervention and at the two and fourth weeks following the intervention.
  Postural Assessment Scale for Stroke is used to assess patients' postural.
Respiratory function | Questionnaire were filled out three times, before the program intervention and at the two and fourth weeks following the intervention.
  Respiratory function was assessed by the technical staff in the rehabilitation ward. examination room
Body awareness | Questionnaire were filled out three times, before the program intervention and at the two and fourth weeks following the intervention.
  Body Awareness Questionnaire is used to assess patients' body awareness.
stroke impact | Questionnaire were filled out three times, before the program intervention and at the two and fourth weeks following the intervention.
  Stroke Impact Scale is used to assess patients' quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang Chu Pai, PhD, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No